CLINICAL TRIAL: NCT04625387
Title: Efficacy of Dry Needle With Exercise In Cervicogenic Headache
Brief Title: Dry Needle In Management of Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raj Nursing and Paramedical College (Other)
Responsible Party: Principal Investigator, Sharick Shamsi, Principal Investigator, Raj Nursing and Paramedical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RajNursingParamedical
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cervicogenic Headache
Keywords: Dry Needle; Exercise; Neck pain; Trigger point
MeSH Terms: conditions — Post-Traumatic Headache; Motor Activity; Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needle plus exercise (Experimental): Group A received Dry Needling along with exercise having 25 individuals. Treatment lasted four weeks duration, twice a week.
  Interventions: Other: Dry Needle and Exercise
- Dry Needling alone (Experimental): Group B received Dry Needling alone having 25 individuals. Treatment lasted four weeks duration, twice a week.
  Interventions: Other: Dry Needle and Exercise

INTERVENTIONS:
Other: Dry Needle and Exercise — A 0.25 X 15 mm acupuncture needle was used for sub occipital muscle and 0.25 X 40 mm needle was used for paraspinal and trapezius muscle. All the necessary precautions were maintained before inserting the needle. Therapists wore hand gloves for all purposes.
  The exercise for the muscles of cervical group, for group A was carried out by elevating head from lying in supine position repeating 20 times in three sets and pressing a theraband forward in one set of 15 repetitions, to right side and to left side and back side
  Other Names: Ice pack

SUMMARY:
Headache is an important health problem. It is the commonest type of all signs of illness in the people worldwide. Cervicogenic Headache is commonest musculoskeletal condition in physiotherapy practice. This study's main objective was to evaluate effectiveness of Dry Needle with exercise in decreasing pain and improving function in patients with Cervicogenic Headache.

DETAILED DESCRIPTION:
50 patients were included and assigned randomly to group A and B. Group-A received Dry Needle plus exercise and group-B received Dry Needle alone. Baseline assessment was taken before and after treatment; treatment was given for four weeks twice a week. Outcome indicators were measured by Visual analog scale, Neck Disability Index and Cervical Range Of Motion.

The study findings indicate that both groups improve the symptoms of a headache. Clinically better improvement was indicated by Dry Needle plus exercise group than Dry Needle alone group. As per our results, Dry Needle plus exercise should be preferred for the management of cervicogenic headache over Dry Needle alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-50 years.
* Male and female both gender
* Worker in the Office.
* Employed permanently.
* Self-motivated for working continuously for rehab.
* Persistent or regular pain in the neck over a span of at least 6 months.

Exclusion Criteria:

* Cervical spine injury or surgery.
* Congenital spinal deformity.
* Participants having age less than 20 or elder than 50 years.
* Cervical radiculopathy,
* The participants had experienced any recent trauma or suffering from dizzy spells, any vascular neurological disorders.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | four weeks
  Visual analogue scale is a subjective outcome measurement where patients judge the intensity of their pain on a scale of 0-10, which is in the form of a 10cm straight line . On this 0-10 scale, zero denotes no pain and ten denotes severe pain intensity
Neck Disability Index | four weeks
  The Neck Disability index contains 10 items, seven related to activities of daily living, two related to pain, and one item related to concentration. Each item is scored ranging from 0 (no pain or disability) to 5 (severe pain and disability); and the total score is expressed as a percentage, with higher scores corresponding to greater disability.

SECONDARY OUTCOMES:
Cervical Range of Motion | four weeks
  Range of motion of cervical spine is being measured by universal goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Sharick Shamsi, PhD, Principal Investigator — Raj Nursing and Paramedical College
Locations (1):
- Sharick Shamsi, Gorakhpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No